CLINICAL TRIAL: NCT04279548
Title: Posterior-superior Insula Deep Brain Stimulation in Refractory Peripheral Neuropathic Pain Patients
Acronym: PSI-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSI-DBS
Record Dates: First submitted 2020-02-04; First posted 2020-02-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Neuropathic Pain; Neuropathy;Peripheral
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Neuralgia; Neuritis | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- On DBS (Active Comparator): Patients in the on mode DBS
  Interventions: Device: Deep Brain Stimulation
- Off DBS (Sham Comparator): Patients in the off mode DBS
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Patients will have a stimulation electrode inserted neurosurgically by neuronavigation to the PSI, on the target used for drTMS, on the insula contralateral to the pain side. After surgery will be randomized to be in in either the ON or OFF DBS

SUMMARY:
This study evaluates the long term pain relief after deep brain stimulation on posterior-superior insula (PSI) in patients with refractory peripheral neuropathic pain who responded to real but not to sham non-invasive stimulation by deep repetitive transcranial magnetic stimulation - PSI-drTMS.

DETAILED DESCRIPTION:
This study has two phases:

Study I) This study is an extension of 690.455/NCT01932905, in which non invasive stimulation of the posterior-superior insula (PSI) was performed by deep repetitive transcranial magnetic stimulation (drTMS) in patients with central neuropathic pain. Patients responding to active stimulation would be invited to join a phase II study aiming at the long term effects of drTMS by deep brain stimulation (DBS) of the PSI. The original 690.455/NCT01932905 study was negative concerning pain intensity reduction compared to sham stimulation, its main outcome. However, in this same study, active but not sham PSI stimulation provided significant anti-nociceptive effects, with anti-allodynic and anti-hyperalgesic properties.

This, and a number of experimental studies on peripheral neuropathic pain relief after PSI stimulation has lead us to perform an extension of the initial study, now including patients with refractory peripheral neuropathic pain to receive an induction series (5 consecutive daily stimulation sessions) of navigated PSI-deep rTMS against sham stimulation in a cross-over design. The calculate sample size for this cross-over screening study is 32. The primary endpoint is number of patients reaching significant pain relief (>50% pain intensity reduction assessed by visual analogue scale (VAS) ranging from 0: no pain, to 100mm:maximal pain imaginable) one week after the 5th stimulation session compared to baseline assessment. Other pain, quality of life and mood data were collected : pain interference with daily living (brief pain inventory), medication quantification score, neuropathic pain symptom inventory (NPSI).

In this screening trial, actual responders: patients refractory peripheral neuropathic pain with >50% pain intensity reduction after real but not sham PSI-drTMS will be offered the opportunity to join a subsequent PSI-DBS phase II trial.

Study II) In this phase, the PSI-DBS phase II trial (ethics review board number #690.455) will enroll 10 patients with refractory peripheral neuropathic pain from study 1 who responded to real but not to sham PSI-drTMS. Patients will have a stimulation electrode inserted neurosurgically by neuronavigation to the PSI, on the target used for drTMS, on the insula contralateral to the pain side.

After surgery, patients will be randomized to be in in either the ON or OFF DBS mode for three months, and then, after a flexible washout period, participants will be switched to the other corresponding mode (OFF or ON) for more three months. The study main outcome is number of responders (number of patients achieving >30% pain intensity reduction). Pain intensity will be measured on a 11-point visual numerical scale anchored at 0 (no pain) and 10 (maximal pain imaginable) and the score at the end of the three-month ON/OFF conditions will be compared to the respective baseline values in order too classify patients as responders or non-responders in each of the ON/OFF conditions. The main secondary outcome is safety, along with other clinical and general patients characteristics such as quality of life( QoL), mood, pain characteristics (McGill Pain Questionnaire-MPQ) and neuropathic pain symptom clusters (Neuropathic Pain Symptom Inventory).

After the ON/OFF double blinded period (main outcome) patients will be maintained for 3 months in the ON mode in a single blinded design, and then for more 6 months, maintained in the open phase of the study. This followup phase will allow us to gain insights into the potential long term effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women aged 21-70 years.
* Ability to give informed consent in accordance with institutional policy.
* Have a diagnosis of neuropathic pain according to Douleur neuropathique 4 questions (DN4).
* Patients with predominant pain on the face and upper extremities in relation to the lower limbs. In this study, predominance will be defined as the difference of ≥ 30% or ≥ 2 points on the VAS scale between upper limb / face pain and lower limb pain.
* Pain lasting more than 12 months.
* Documented resistance to clinical treatment, defined in this study as persistence of pain after a minimum of 2 appropriate pharmacological treatments, including at least one antidepressant / anticonvulsant and / or gabapentins. Adequacy of treatments will be defined by the use of drugs in doses considered adequate in the literature or below the threshold of side effects.
* Visual analog scale (EVA) scores of at least four during initial assessments.
* No change in the analgesic medication regimen for chronic neuropathic pain during the 4 weeks preceding entry into the study.
* Ability to comply with the tests and follow-up defined by the study protocol;
* Absence of routine contraindications to the surgical procedure (eg Coagulopathies, blood dyscrasias). These will be evaluated by members of the neurosurgical team responsible for the study

Exclusion Criteria:

* Alcohol abuse, medication, or addiction to illicit substances in the last 12 months.
* Diagnosis of idiopathic trigeminal neuralgia or atypical facial pain.
* Advanced cardiovascular disease stage that makes anesthesia and surgery unsafe, as determined by the neurosurgeon / clinical team.
* Clinically relevant lesions (tumor, for example) on preoperative magnetic resonance imaging.
* Cardiac pacemaker / implanted defibrillator or other active stimulators.
* Medical condition that requires repeated resonances.
* Patients using chemotherapy for the treatment of malignant tumors or who need chronic oral or intravenous treatment with immunosuppressants or steroids.
* Patients unable to comply with the study visit schedule.
* Brain ablative surgery or previous neurosurgery that prevents or increases the risk of implantation of the electrodes.
* Patients of childbearing potential or infants with a positive pregnancy test or without the use of adequate contraception.
* Other medical conditions that require probable hospitalization during the study.
* History of epilepsy or status epilepticus.
* Chronic infection.
* Diagnosis of fibromyalgia.
* Plans for using diathermy in the future.
* Have any intracranial metal implant
* Current participation in another device investigation study or experimentation with drugs or surgery of any kind.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Response (>30% pain intensity reduction) after ON but not OFF stimulation periods. | after 3 months in the ON / OFF conditions
  Pain intensity measured on a Numeric Rating Scale (0-10) where 0 is no pain and 10 is the worst pain imaginable

SECONDARY OUTCOMES:
% of patients with anxiety and depression | baseline, 3 months and 15 months after the intervention
  Assessment of the anxiety and depression by Hospital Anxiety And Depression Scale. The possible scores ranged from 0 to 21 for anxiety and depression. 0 to 7 could be regarded as being in the normal range, a score of 11 or higher indicating probable presence of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state.
Incidence of symptoms of neuropathic pain | baseline, 3 months and 15 months after the intervention
  Symptoms of neuropathic pain evaluated by Neuropathic Pain Symptom Inventory

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by self reported | baseline, 3 months and 15 months after the intervention
  Assessment of adverse events by self-report
Quality of life related to pain relief | baseline, 3 months and 15 months after the intervention
  Quality of life evaluated by WHOQOL-BREF

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participant data for primary and secondary outcome measures will be made available only when requested according with local ethics review recommendations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion

REFERENCES:
- [Derived] Dongyang L, Cunha PHM, Lapa JDS, Kubota GT, Junior JR, Fernandes AM, Thibes RB, Pinheiro DS, Iglesio RF, Duarte KP, Sato J, da Silva VA, Lucato LT, Figueiredo EG, Carlotti Junior CG, Yeng LT, Teixeira MJ, de Andrade DC. Insula Deep Brain Stimulation for Neuropathic Pain: A Cross-Over, Randomized, Sham-Controlled Trial. Neuromodulation. 2025 Aug 18:S1094-7159(25)00261-2. doi: 10.1016/j.neurom.2025.07.001. Online ahead of print. PMID 40824225